CLINICAL TRIAL: NCT02011321
Title: Clevidipine for Vasospasm After Subarachnoid Hemorrhage
Brief Title: Clevidipine for Vasospasm After Subarachnoid Hemorrhage (SAH)
Acronym: CLEVAS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Panayiotis Varelas, Division Head Neurosciences Critical Care, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HFHS-CLEVIDIPINE-PV
Record Dates: First submitted 2013-12-02; First posted 2013-12-13 (Estimated); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Subarachnoid Hemorrhage; Cerebral Aneurysm; Vasospasm, Intracranial
Keywords: subarachnoid hemorrhage; aneurysm; vasospasm; clevidipine; transcranial dopplers
MeSH Terms: conditions — Subarachnoid Hemorrhage; Intracranial Aneurysm; Vasospasm, Intracranial; Aneurysm | interventions — clevidipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- clevidipine (Experimental): Four-hour infusion of low-dose intravenous clevidipine in patients with moderate vasospasm after aneurysmal subarachnoid hemorrhage
  Interventions: Drug: clevidipine

INTERVENTIONS:
Drug: clevidipine — clevidipine infusion x4 hours
  Other Names: Cleviprex

SUMMARY:
Vasospasm occurs frequently after aneurysmal subarachnoid hemorrhage and can lead to strokes. The investigators will investigate if infusion of a novel drug, clevidipine, will decrease vasospasm during the infusion and post infusion period using transcranial doppler monitoring of patients with subarachnoid hemorrhage and moderate severity vasospasm

DETAILED DESCRIPTION:
Cerebral vasospasm after aneurysmal subarachnoid hemorrhage (SAH) is a major cause of morbidity and mortality days after securing the aneurysm due to development of cerebral ischemia and strokes. Vasospasm is detected by measuring the blood flow velocities in the cerebral circulation via daily Transcranial Dopplers (TCD). There is no effective treatment except for a per os calcium channel blocker (nimodipine) and for keeping the patient hypertensive and with euvolemia or hypervolemia. A recently proposed option is to dilate the cerebral vessels by infusing continuously another vasodilatory calcium channel blocker, nicardipine, and supporting the systemic blood pressure (BP) with vasopressors which do not constrict the cerebral vasculature at the same time. Nicardipine has also been used extensively intra-arterially as a bolus or infusion to dilate the vasospastic cerebral vessels as a rescue therapy for severe vasospasm.

Clevidipine is a novel, short-acting calcium channel blocker, which in a small series of patients with SAH at Henry Ford Hospital, was able to control the elevated BP very efficiently and within a narrow window, without adverse events. It has never been used before for ameliorating vasospasm, but theoretically offers advantages compared to nicardipine due to its shorter half-life and easier titratability. Except for use of clevidipine for BP control in the investigators previous study, there are no data on clevidipine use after SAH and no data about effect of the drug on vasospasm.

In this single-center, open-label, uncontrolled, pilot clinical study, the investigators hypothesize that clevidipine low-rate infusion will decrease sonographically-detected moderate cerebral vasospasm after aneurysmal SAH. The dose of the drug in this exploratory study is 2.5 to 5 times lower than the dose used previously to control BP. The effect of the drug will be evaluated in 20 patients by TCD monitoring during 3 periods: 1-hour pre-infusion, 4-hour infusion and 4-hour post infusion. The cerebral blood flow velocities, which are a surrogate marker of vasospasm, will be compared between the 3 periods. The primary efficacy end-point will be the percentage of measurements with at least a 10% or more decrease of the velocities during the infusion period. Potential long-term effects after discontinuation of the drug will be also evaluated in the post-infusion 4-hour period and beyond, until the last follow up. The major safety issue is hypotension induced by the drug during a period when vasospasm is present. For that reason, two measures will be taken. First, only patients with moderate vasospasm will be evaluated. Second, vasopressors will be used as needed during the infusion period to counteract the systemic circulatory effect of the drug and maintain a stable systemic Mean Arterial Pressure (MAP) within 10% range compared to pre-infusion. Potential effect of cerebral vasodilation on intracranial pressure (ICP) will be also evaluated during the infusion and post-infusion periods and any elevation > 10 mm Hg will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Diagnosis of SAH (as diagnosed per history, neuroimaging or lumbar puncture)
* Presence of a secured aneurysm via clipping or coiling
* Hunt and Hess grade < 5 (non-sedated or paralyzed patients)
* Glasgow Coma scale > 4 (non-sedated or paralyzed patients)
* MAP goal set by the treating physicians
* Temporal insonation window presence on TCD
* Moderate supratentorial vasospasm as per daily TCD (CBFV between 130-180 cm/sec or Lindergaard index 3-5 for the Middle Cerebral artery or Internal Cerebral artery or Anterior Cerebral artery)

Exclusion Criteria:

* Very young or very old patients (<18 or >80 years old)
* Traumatic SAH (no aneurysm identified after initial work-up) or Perimesencephalic SAH is also excluded
* Hunt and Hess grade 5 (deeply comatose or brain dead patients)
* Glasgow Coma scale 3 or 4 (brain dead or deeply comatose patients)
* Patients with mild or severe supratentorial vasospasm (CBFV < 120 cm/sec or Lindergaard index < 3 or > 200 cm/sec or Lindergaard index > 6, respectively, for the Middle Cerebral artery or Internal Cerebral artery or Anterior Cerebral artery)
* Patients with vasospasm only in the posterior circulation (CBFV > 80 cm/sec for Vertebral or Basilar artery)
* Patients with severe tachycardia (heart rate > 110)
* Patients with preexisting left bundle branch block or permanent ventricular pacemaker
* Patients with known allergy to dihydropyridines including clevidipine or allergic to soybeans, soy products, eggs, or egg products
* Patients with defective lipid metabolism such as pathologic hyperlipemia or lipoid nephrosis
* Patients with acute pancreatitis, if it is accompanied by hyperlipidemia
* Patients with severe aortic stenosis
* Pregnant patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2018-03 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Change of cerebral blood flow velocities during infusion of clevidipine compared to baseline pre-infusion by >10% at 15 min after start of infusion and/or at 1, 2,3 and 4 hours (during the infusion). | 15 min after start of infusion and at 1, 2,3 and 4 hours (during the infusion).
  Efficacy: We will compare pre-infusion, infusion and post-infusion CBFVs measured by TCD as a surrogate of vasospasm. We will assess the percentage of measurements meeting the primary outcome of 10% change of cerebral blood flow velocities during the infusion period compared to pre-infusion

SECONDARY OUTCOMES:
Safety and Tolerability: Intracranial pressure (ICP) change during infusion compared to pre-infusion | ICP will be measured at the end of pre-infusion period and at the end of the infusion period
  The mean difference between pre-infusion and end-of-infusion ICP will be calculated. Any change > 10 mm Hg (elevation or decrease) will be reported as a safety issue
Safety and tolerability: pressor requirement to counteract a 10% or more drop of mean arterial pressure (MAP) during the infusion period | MAP measurements every minute during the pre-infusion and infusion period
  Safety & Tolerability: if during infusion the Mean arterial pressure drops > 10% compared to pre-infusion (mean MAP measurements during this period), a pressor (neosynephrine) drip will be initiated to counteract this effect systemically and bring the MAP at the mean pre-infusion level. The percentage of participants who will need this rescue treatment will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Panayiots Varelas, MD, PhD, Principal Investigator — Henry Ford Health System; Tamer Abdelhak, MD, Study Director — Henry Ford Health System; Mohammed Rehman, DO, Study Director — Henry Ford Health System
Locations (1):
- Henry Ford hospital, Detroit, Michigan, United States

REFERENCES:
- [Background] Varelas PN, Abdelhak T, Corry JJ, James E, Rehman MF, Schultz L, Mays-Wilson K, Mitsias P. Clevidipine for acute hypertension in patients with subarachnoid hemorrhage: a pilot study. Int J Neurosci. 2014 Mar;124(3):192-8. doi: 10.3109/00207454.2013.836703. Epub 2013 Sep 24. PMID 24007334
- [Background] Espina IM, Varon J. Clevidipine : a state-of-the-art antihypertensive drug under the scope. Expert Opin Pharmacother. 2012 Feb;13(3):387-93. doi: 10.1517/14656566.2012.651126. Epub 2012 Jan 18. PMID 22251017
- See also: Clevidipine information — http://www.cleviprex.com/